CLINICAL TRIAL: NCT06315933
Title: Long-term Effect of General Anesthesia Before School Age on Neurodevelopment in Children With Congenital Scoliosis
Brief Title: Anesthesia Neurodevelopmental Impact in Congenital Scoliosis Children
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lulu Ma, Chief physician, Professor, Peking Union Medical College Hospital
Other Study IDs: S-K1093
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: General Anesthetics Toxicity
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unexposed: Children unexposed to general anesthesia before school age (<=6y)
- Singly exposed: Children singly exposed to general anesthesia before school age (<=6y)
  Interventions: Procedure: General anesthesia
- Multiply exposed: Children multiply exposed to general anesthesia before school age (<=6y)
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: General anesthesia — General anesthesia including inhaled and intravenous
  Groups: Multiply exposed; Singly exposed

SUMMARY:
In the past, a large number of animal studies have suggested that anesthesia exposure has potential neurotoxic effects, resulting in persistent cognitive and behavioral deficits. At present, there is still a lack of sufficient clinical research evidence to prove whether anesthesia exposure has long-term effects on neurodevelopment. The existing clinical research data suggests that a single short-time anesthesia exposure in young children does not affect long-term neurodevelopmental outcomes. Early onset scoliosis, including congenital scoliosis, is a type of scoliosis deformity that occurs before the age of 10. Posterior scoliosis correction surgery is one of the common treatment. There is currently no research indicating the impact of early single or multiple long-duration anesthesia exposure on the neurological development of children with congenital scoliosis. The aim of this study is to determine the long-term effect of general anesthesia exposure on neurocognitive function and behavior in children with congenital scoliosis, in order to provide reference for related clinical work.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital scoliosis
* 6-16 years old at the time of assessment

Exclusion Criteria:

* Cognitive impairment caused by congenital, traumatic or other reasons;
* Existence of mental or psychological disorders;
* There are factors that may affect neurological development, including any known central nervous system disease, neurological injury, or history of neonatal asphyxia;
* Unable to cooperate with cognitive function tests;
* The child is unable to communicate in Chinese.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with congenital scoliosis
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
full-scale intelligence quotient, FSIQ | At the time of collecting baseline demographic data
  Measured by Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV)

SECONDARY OUTCOMES:
Verbal Comprehension Index (VCI), Perceptual Reasoning/Organization Index (PRI/POI) | At the time of collecting baseline demographic data
  Measured by Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV)
CBCL Total score, CBCL Internalizing score, CBCL Externalizing score | Within six months of WISC-IV assessment
  Measured by Child Behavior Checklist (CBCL)
SDQ total difficulties score, SDQ internalizing problems score, SDQ externalizing problems score, SDQ prosocial behavior score | Within six months of WISC-IV assessment
  Measured by Strengths and Difficulties Questionnaire (SDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Lulu Ma, Dr., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 1 year after the results are published
Access Criteria: IPD is available on appropriate request from the Principle Investigator by email

REFERENCES:
- [Background] Istaphanous GK, Ward CG, Nan X, Hughes EA, McCann JC, McAuliffe JJ, Danzer SC, Loepke AW. Characterization and quantification of isoflurane-induced developmental apoptotic cell death in mouse cerebral cortex. Anesth Analg. 2013 Apr;116(4):845-54. doi: 10.1213/ANE.0b013e318281e988. Epub 2013 Mar 4. PMID 23460572
- [Background] Brambrink AM, Back SA, Riddle A, Gong X, Moravec MD, Dissen GA, Creeley CE, Dikranian KT, Olney JW. Isoflurane-induced apoptosis of oligodendrocytes in the neonatal primate brain. Ann Neurol. 2012 Oct;72(4):525-35. doi: 10.1002/ana.23652. PMID 23109147
- [Background] Briner A, De Roo M, Dayer A, Muller D, Habre W, Vutskits L. Volatile anesthetics rapidly increase dendritic spine density in the rat medial prefrontal cortex during synaptogenesis. Anesthesiology. 2010 Mar;112(3):546-56. doi: 10.1097/ALN.0b013e3181cd7942. PMID 20124985
- [Background] Zhang H, Du L, Du Z, Jiang H, Han D, Li Q. Association between childhood exposure to single general anesthesia and neurodevelopment: a systematic review and meta-analysis of cohort study. J Anesth. 2015 Oct;29(5):749-57. doi: 10.1007/s00540-015-2030-z. Epub 2015 May 23. PMID 26002228
- [Background] McCann ME, de Graaff JC, Dorris L, Disma N, Withington D, Bell G, Grobler A, Stargatt R, Hunt RW, Sheppard SJ, Marmor J, Giribaldi G, Bellinger DC, Hartmann PL, Hardy P, Frawley G, Izzo F, von Ungern Sternberg BS, Lynn A, Wilton N, Mueller M, Polaner DM, Absalom AR, Szmuk P, Morton N, Berde C, Soriano S, Davidson AJ; GAS Consortium. Neurodevelopmental outcome at 5 years of age after general anaesthesia or awake-regional anaesthesia in infancy (GAS): an international, multicentre, randomised, controlled equivalence trial. Lancet. 2019 Feb 16;393(10172):664-677. doi: 10.1016/S0140-6736(18)32485-1. Epub 2019 Feb 14. PMID 30782342
- [Background] Zaccariello MJ, Frank RD, Lee M, Kirsch AC, Schroeder DR, Hanson AC, Schulte PJ, Wilder RT, Sprung J, Katusic SK, Flick RP, Warner DO. Patterns of neuropsychological changes after general anaesthesia in young children: secondary analysis of the Mayo Anesthesia Safety in Kids study. Br J Anaesth. 2019 May;122(5):671-681. doi: 10.1016/j.bja.2019.01.022. PMID 30982593
- [Background] Baky FJ, Milbrandt TA, Flick R, Larson AN. Cumulative Anesthesia Exposure in Patients Treated for Early-Onset Scoliosis. Spine Deform. 2018 Nov-Dec;6(6):781-786. doi: 10.1016/j.jspd.2018.05.001. PMID 30348358
- [Background] Ruiz G, Torres-Lugo NJ, Marrero-Ortiz P, Guzman H, Olivella G, Ramirez N. Early-onset scoliosis: a narrative review. EFORT Open Rev. 2022 Aug 4;7(8):599-610. doi: 10.1530/EOR-22-0040. PMID 35924646
- [Background] Zhang Q, Peng Y, Wang Y. Long-duration general anesthesia influences the intelligence of school age children. BMC Anesthesiol. 2017 Dec 19;17(1):170. doi: 10.1186/s12871-017-0462-8. PMID 29258430
- [Background] Lin T, Meng Y, Ji Z, Jiang H, Shao W, Gao R, Zhou X. Extent of Depression in Juvenile and Adolescent Patients with Idiopathic Scoliosis During Treatment with Braces. World Neurosurg. 2019 Jun;126:e27-e32. doi: 10.1016/j.wneu.2019.01.095. Epub 2019 Jan 29. PMID 30703588
- [Derived] Dai Z, Zhang Y, Ma L, Zhang J, Huang Y. Association between general anaesthesia exposure and neurodevelopment in children with congenital scoliosis at a Chinese tertiary hospital: study protocol for a prospective longitudinal observational cohort study. BMJ Open. 2025 Dec 2;15(12):e108845. doi: 10.1136/bmjopen-2025-108845. PMID 41338617